CLINICAL TRIAL: NCT06147453
Title: Effect of the Aerobika Oscillating Positive Expiratory Pressure (OPEP) Device on Mucus Plugging and Airflow Obstruction in Patients with Moderate-to-severe Asthma
Brief Title: Effect of OPEP on Mucus Plugging and Airflow Obstruction in Patients with Moderate-to-severe Asthma
Acronym: AeroMUC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Trudell Medical International (Industry)
Responsible Party: Principal Investigator, Sarah Svenningsen, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIRH-Xe011
Record Dates: First submitted 2023-11-15; First posted 2023-11-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Aerobika OPEP device (Active Comparator): The OPEP system (Aerobika®) combines positive expiratory pressure therapy and airway vibrations to help mobilize pulmonary secretions. OPEP therapy (Aerobika ®) enforces resistance to exhalation at the mouth, while the airway vibration technology transmits movements upstream during exhalation so that airway walls may become free from mucus.
  Participants will take home the device and use it twice daily for 16 weeks.
  Interventions: Device: Aerobika OPEP device
- Standard of care (No Intervention): Standard of care management for 16 weeks.

INTERVENTIONS:
Device: Aerobika OPEP device — 16 week twice daily use of the Aerobika OPEP device
  Arms: Aerobika OPEP device

SUMMARY:
The goal of this randomized clinical trial is to evaluate the effect of daily AerobikaTM Oscillating Positive Expiratory Pressure (OPEP) device use on mucus plugging and airway function in adult patients with moderate-to-severe asthma.

DETAILED DESCRIPTION:
Airway mucus occlusions have been identified as an important feature of asthma pathophysiology. The use of an airway clearance device may help clear such mucus plugs and consequently improve airway function and asthma control. Therefore, we will investigate the effects of daily Aerobika Oscillating Positive Expiratory Pressure (OPEP) device use in a two-centre, randomized, open-label study of adult patients with moderate-to-severe asthma that is uncontrolled with evidence of mucus plugging.

The total study duration per patient will be 17 weeks, consisting of a screening period of up-to 1 week, and an open-label randomized treatment period of 16 weeks. Participants will be randomized to Aerobika use or will continue their current medications. The trial will evaluate the effect of Aerobika use on mucus plugging, airway function, and asthma control.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent.
2. Able and willing to comply with the study protocol.
3. Males and females ≥ 18 years of age.
4. Asthma diagnosed by a respiratory physician ≥12 months prior to study enrolment based on the Global Initiative for Asthma (GINA) 2014 guidelines - GINA 4 or 5.
5. ICS dose ≥500 mcg of fluticasone equivalent/day. Patients on prednisone or biologic for ≥3 months would not be excluded as long as they meet the rest of the inclusion criteria.
6. ACQ ≥1.5 during the screening period.
7. CT mucus score ≥4 during the screening period.

Exclusion Criteria:

1. Acute or chronic parasitic, bacterial, fungal or viral infections that required, or currently requires, hospitalization or antimicrobial treatment during the last four weeks.
2. Acute asthma exacerbation event treated with increased doses of oral, or any dose of intramuscular (IM) or intravenous (IV) corticosteroids within six weeks prior to screening.
3. Other relevant pulmonary diseases (e.g., chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, cystic fibrosis, pulmonary arterial hypertension, tuberculosis) requiring treatment within 12 months prior to screening.
4. Alcohol or substance abuse within 12 months prior to screening.
5. Current smoker defined as having smoked at least one cigarette (or pipe, cigar, or cannabis) per day for ≥ 30 days within the three months prior to screening.
6. Ex-smokers with ≥ 15 pack-year smoking history.
7. Patient has an implanted mechanically, electrically, or magnetically activated device or any metal in their body which cannot be removed, including but not limited to pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures and/or ear implants) (at the discretion of the MRI Technologist).
8. In the investigator's opinion, subject suffers from any physical, psychological, or other condition(s) that might prevent performance of the MRI, such as severe claustrophobia.
9. Pregnant or breastfeeding
10. Participation in any clinical trial of an investigational agent or procedure within three months prior to screening or during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Computed Tomography (CT) mucus score | 16 weeks
  Change in the CT mucus score between screening/baseline (week 0) and week 16. Mucus scores range from 0 (best outcome) to 20 (worst outcome).

SECONDARY OUTCOMES:
MRI ventilation defect percent (VDP) | 16 weeks
  Change in MRI VDP between screening/baseline (week 0) and week 16.
Forced expiratory volume in one second (FEV1) | 16 weeks
  Change in FEV1 between screening/baseline (week 0) and week 16.
Asthma Control Questionnaire-5 (ACQ-5) | 16 weeks
  Change in ACQ-5 between screening/baseline (week 0) and week 16. ACQ-5 ranges from 0 (best outcome) to 5 (worst outcome).
Asthma Quality of Life Questionnaire (AQLQ) | 16 weeks
  Change in AQLQ between screening/baseline (week 0) and week 16. AQLQ ranges from 1 (worst outcome) to 7 (best outcome).
Asthma Control Test (ACT) | 16 weeks
  Change in ACT between screening/baseline (week 0) and week 16. ACT ranges from 5 (worst outcome) to 25 (best outcome).
Cough and Sputum Assessment Questionnaire (CASA-Q) | 16 weeks
  Change in CASA-Q between screening/baseline (week 0) and week 16. The scores for each domain range from 0 to 100, with higher scores indicating fewer/less severe symptoms and less impact.
St. George's Respiratory Questionnaire (SGRQ) | 16 weeks
  Change in SGRQ between screening/baseline (week 0) and week 16. SGRQ scores range from 0 to 100, with higher scores indicating more limitations.
fraction of exhaled nitric oxide (FeNO) | 16 weeks
  Change in FeNO between screening/baseline (week 0) and week 16.
blood eosinophil count | 16 weeks
  Change in blood eosinophil count between screening/baseline (week 0) and week 16.
sputum eosinophil percent | 16 weeks
  Change in sputum eosinophil percent between screening/baseline (week 0) and week 16.
sputum neutrophil percent | 16 weeks
  Change in sputum neutrophil percent between screening/baseline (week 0) and week 16.
inspiratory CT wall area percent (WA%) | 16 weeks
  Change in CT WA% between screening/baseline (week 0) and week 16.
inspiratory CT lumen area (LA) | 16 weeks
  Change in CT LA between screening/baseline (week 0) and week 16.
respiratory system resistance (Rrs) at 5Hz | 16 weeks
  Change in Rrs5Hz between screening/baseline (week 0) and week 16.
respiratory system reactance (Xrs) at 5Hz | 16 weeks
  Change in Xrs5Hz between screening/baseline (week 0) and week 16.
respiratory system resistance (Rrs) at 19Hz | 16 weeks
  Change in Rrs19Hz between screening/baseline (week 0) and week 16.
frequency dependence of Rrs (Rrs5-19Hz) | 16 weeks
  Change in Rrs5-19Hz between screening/baseline (week 0) and week 16.
integrated area of low frequency reactance (AX) | 16 weeks
  Change in AX between screening/baseline (week 0) and week 16.

OTHER OUTCOMES:
Sputum rheology | 16 weeks
  Change from screening/baseline (week 0) to week 16 in expectorated sputum rheology (critical stress, elastic modulus, viscous modules)
Mucin proteins in sputum | 16 weeks
  Change from screening/baseline (week 0) to week 16 in mucin proteins in sputum (MUAC5, MUCSB, MUC5AC:MUC5B ratio).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Western University, London, Ontario

IPD SHARING:
Plan to Share IPD: No